CLINICAL TRIAL: NCT06834672
Title: A Multicenter, Randomized, Open-label Phase III Study of IBI354 Versus Investigator's Choice of Chemotherapy in Patients With Platinum-resistant Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Brief Title: Study of IBI354 Versus Investigator's Choice of Chemotherapy in Patients With Platinum-resistant Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CIBI354A301
Record Dates: First submitted 2025-02-05; First posted 2025-02-19 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Ovarian; Primary Peritoneal; Fallopian Tube Cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm, Control Arm (Experimental)
  Interventions: Drug: IBI354
- Control drug (Active Comparator)
  Interventions: Drug: paclitaxel/Gemcitabine/Liposomal doxorubicin

INTERVENTIONS:
Drug: IBI354 — intravenous infusion of 12 mg/kg on Day 1 of each 3-week treatment cycle
  Arms: Experimental Arm, Control Arm
Drug: paclitaxel/Gemcitabine/Liposomal doxorubicin — paclitaxel：- Usage and dosage: 80 mg/m2 administered as an intravenous infusion on Day 1 of each weekly treatment cycle。 Gemcitabine：Usage and dosage: intravenous infusion at 1000 mg/m2 on Days 1, 8 of each 3-week treatment cycle。 Liposomal doxorubicin：Usage and dosage: intravenous infusion of 40 mg/m2 on Day 1 of each 4-week treatment cycle
  Arms: Control drug

SUMMARY:
This is a multiregional, multicenter, randomized, open-label, phase III study to compare the efficacy, safety, and tolerability of IBI354 monotherapy with investigator's choice of chemotherapy (paclitaxel, gemcitabine, liposomal doxorubicin, or topotecan) in patients with HER2-expressing, platinum-resistant ovarian, primary peritoneal, or fallopian tube cancer.

Participants with advanced ovarian, primary peritoneal, fallopian tube cancer who have failed or are intolerant to first-line or more platinum-based chemotherapy will be randomly assigned in a 2:1 ratio to two treatment arms:

Experimental Arm: IBI354 monotherapy arm, 12 mg/kg IBI354 on Day 1 of each 3-week cycle; Control Arm: Investigator's choice chemotherapy (paclitaxel, gemcitabine, liposomal doxorubicin, or topotecan)

ELIGIBILITY:
Inclusion Criteria

1. Participants have the ability to understand and give written informed consent Form (ICF) for participation in this trial, including all evaluations and procedures as specified by this protocol;
2. Female participants ≥ 18 years old;
3. Expected life time ≥ 12 weeks
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
5. Histologically or cytologically confirmed locally advanced unresectable or metastatic ovarian, primary peritoneal, or fallopian tube cancer.
6. Must have confirmed disease progression during or after the most recent anticancer therapy.
7. Must have at least 1 measurable target lesion per RECIST v1.1 criteria.
8. Left Ventricular Ejection Fraction (LVEF) ≥ 50% within 28 days prior to the first dose of study drug.
9. Adequate bone marrow and organ function.
10. Female participants of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of study drug and use effective contraception throughout the treatment period and for 6 months after the treatment period.

Exclusion Criteria:

1. Patients with histological or cytological findings meet any of the following criteria:

   1. Endometrioid tumor, clear cell tumor, mucinous tumor, mesenchymal tumor, or contains any of the above components.
   2. Low-grade or borderline tumor, or contains any of the above components.
2. Participation in any other interventional clinical study, except observational (non-interventional) study.
3. Paclitaxel, gemcitabine, liposomal doxorubicin, and topotecan listed in the control arm were either ineligible or had previously received and progressed.
4. Prior therapy to first dose of study drug:

   1. Participants who have been treated with Intravenous infusion of chemotherapeutic drugs, macromolecular targeted drugs, immunotherapy, intraperitoneal chemotherapy, tumor embolization or interventional chemotherapy, within 4 weeks.
   2. Participants who have been treated with oral chemotherapeutic drugs, small molecular targeted drugs, endocrine therapy, and Chinese herbal medicine for anticancer treatment indications, within 2 weeks or 5 half-lives (whichever is longer).
   3. Participants who have been treated with radical radiotherapy within 4 weeks, palliative radiotherapy within 2 weeks.
   4. Participants who have been treated with strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers within 2 weeks or 5 half-lives (whichever is longer).
   5. Participants who have been treated with Major surgery (craniotomy, thoracotomy or laparotomy and other types of surgery considered "major" by the investigator, excluding needle biopsy) within 4 weeks; Laparoscopic exploration surgery within 2 weeks. Or participants have serious non-healing wound, trauma or ulcer.
   6. Participants who have been treated with live vaccines (mRNA and non-replicating adenovirus vaccines are not considered live vaccines) within 4 weeks.
5. Have adverse reactions caused by previous anti-tumor therapy that have not been resolved to Grade 0 or 1 according to NCI-CTCAE v5.0 criteria.
6. Presence of symptomatic central nervous system (CNS) metastases, spinal cord compression, carcinomatous meningitis, or history of leptomeningeal carcinoma.
7. Participants with pneumonitis requiring corticosteroid treatment, or a history of other clinically significant lung disease.
8. Uncontrolled or significant cardiovascular and cerebrovascular disease.
9. Use of immunosuppressive medications within 14 days prior to the first dose of study treatment.
10. Tumor invades surrounding important tissues or organs.
11. Bleeding within 3 months prior to the first dose of study treatment.
12. Symptomatic abdominal or pelvic effusion requiring intervention.
13. Esophageal or gastric varices that require immediate intervention (e.g., ligation or sclerotherapy), or have high risk of bleeding considered by the investigator or gastroenterology and hepatology specialists; participants with evidence of portal hypertension.
14. Unhealed gastrointestinal obstruction, perforation, or fistula, or participants at risk for gastrointestinal obstruction or perforation.
15. Have intraluminal stenting of the digestive tract or trachea.
16. Participants with biliary obstruction will be excluded.
17. Participants with hepatic encephalopathy, hepatorenal syndrome, or cirrhosis of Child-Pugh class B or above.
18. Significant malnutrition.
19. Uncontrolled active infection.
20. Concomitant other primary malignancies within 3 years or other malignancies with active or risk of recurrence before the first dose of study treatment.
21. History of immunodeficiency disease, including congenital or acquired immunodeficiency disease.
22. History of allogeneic organ transplantation, allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation.
23. Allergy to other anti-HER2 antibodies/ADC or any component of IBI354.
24. Participants who are pregnant or lactating, or those who plan to become pregnant.
25. Other acute or chronic diseases or laboratory abnormalities that may increase the risk of participation in the study or administration of the study treatment, interfere with the interpretation of the study results, or lead the investigator to determine that the participant is inappropriate for participation in the study.
26. The participant has neurological, psychiatric, or social conditions that affect trial compliance, significantly increase the risk of adverse events, or affect the participant's ability to provide written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-12-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
To compare the Progression-free survival (PFS) of IBI354 monotherapy versus investigator's choice of chemotherapy | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
  PFS as evaluated per the RECIST v1.1 criteria
Overall Survival (OS) | From date of randomization until the date of death from any cause (up to approximately 48 months)
  Overall survival

SECONDARY OUTCOMES:
Number of subjects with clinically significant changes in physical examination results | up to approximately 36 months
Numbers of subjects with adverse events | up to approximately 36 months
CA-125 response rate according to Gynecologic Cancer Intergroup (GCIG) criteria. | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
To compare the objective response rate (ORR) of IBI354 monotherapy versus investigator's choice of chemotherapy | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
  ORR as evaluated per the RECIST v1.1 criteria
Disease Control Rate (DCR) of IBI354 monotherapy versus investigator's choice of chemotherapy | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
  DCR as evaluated per the RECIST v1.1 criteria
Duration of Response (DoR) of IBI354 monotherapy versus investigator's choice of chemotherapy | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
  DoR as evaluated per the RECIST v1.1 criteria
Time to Response (TTR) of IBI354 monotherapy versus investigator's choice of chemotherapy | From date of randomization until the occurrence of first documented progression, death from any cause, or the initiation of new anticancer treatment, whichever occurs first (up to approximately 36 months)
  TTR as evaluated per the RECIST v1.1 criteria
Numbers of subjects with adverse Event of Special Interest | up to approximately 36 months
Numbers of subjects with Serious Adverse Event (SAE) | up to approximately 36 months
Evaluate participant's global health status | up to approximately 36 months
  Evaluate participant's global health status by Quality of Life-5 Dimension-5 Level (EQ-5D-5L)
Evaluate participant's cancer-related symptoms and quality of life | up to approximately 36 months
  Evaluate participant's cancer-related symptoms and quality of life by European by Organization for Research and Treatment of Cancer (EORTC) Core Quality of Life Questionnaire-Core 30 (QLQ-C30)
Evaluate the impact of ovarian cancer on participant's physiological, emotional, and social aspects | up to approximately 36 months
  Evaluate the impact of ovarian cancer on participant's physiological, emotional, and social aspects by EORTC Quality of Life Questionnaire-Ovarian Cancer 28 (QLQ-OV28)
Pharmacokinetic (PK) paramenter of IBI354: Plasma concentration (Cmax) | up to approximately 36 months
  Evaluation of the plasma concentration (Cmax) in subjects treated with IBI354
PK paramenter of IBI354: Area under the curve (AUC) | up to approximately 36 months
  Evaluation of the Area under the curve (AUC) in subjects treated with IBI354
PK paramenter of IBI354: Time to maximum concentration (Tmax) | up to approximately 36 months
  Evaluation of the Time to maximum concentration (Tmax) in subjects treated with IBI354
PK paramenter of IBI354: Clearance (CL) | up to approximately 36 months
  Evaluation of the Clearance (CL) in subjects treated with IBI354
PK paramenter of IBI354: Volume of distribution (V) | up to approximately 36 months
  Evaluation of the Volume of distribution (V) in subjects treated with IBI354
PK paramenter of IBI354: Half-life (T1/2) | up to approximately 36 months
  Evaluation of the Half-life (T1/2) in subjects treated with IBI354
Immunogenicity of IBI354: the incidence of anti-drug Antibody(ADA) | up to approximately 36 months
  The proportion of evaluable subjects (those with both baseline and post-baseline ADA measurements) who tested positive for anti-drug antibodies.
Immunogenicity of IBI354: the incidence of Neutralizing Antibody (Nab) (if applicable) | up to approximately 36 months
  The proportion of evaluable subjects (those with both baseline and post-baseline ADA measurements) who tested positive for neutralizing antibodies.
Effect of ADA on safety (if applicable) | up to approximately 36 months
  Assessment of the potential impact of ADA on safety by comparing the incidence of treatment-emergent adverse events (e.g., TEAEs) between ADA-positive and ADA-negative groups.
Effect of ADA on efficacy (if applicable) | up to approximately 36 months
  Assessment of the potential impact of ADA on drug efficacy by comparing primary efficacy endpoints (e.g., PFS, OS) between ADA-positive and ADA-negative groups.
Effect of ADA on PK parameters (if applicable) | up to approximately 36 months
  Assessment of the potential impact of ADA on the PK parameters of IBI354 between ADA-positive and ADA-negative groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Cancer Hospital of Chongqing University, Chongqing, Chongqing Municipality, China